CLINICAL TRIAL: NCT06701435
Title: The Effect of Post-Training Cold Compression on Muscle Oxygen Saturation and Jumping Performance in Professional Men Volleyball Players
Brief Title: The Effect of Post-Training Cold Compression in Professional Volleyball Players
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Seval Tamer, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: KSHU-ST-01
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-10

CONDITIONS: Healthy Men
Keywords: Oxygen saturation; jumping; volleyball; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 Degree Cold Compression Group: Cold compression application was performed using Game Ready for 15 minutes. The target temperature was manually set to 1°C and the pressure was set to high compression (75 mm Hg). Since it is known that the applied pressure increases the effect of cold application and oxygenation in the tissue increases as the compression intensity increases (108), it was applied in the high option. Duration was preferred because the optimal range for the duration of cold applications is given as 11-15 minutes in the literature (120). Pneumatic intermittent compression with a standard ∼3-minute cycle was applied to both lower legs using a thigh wrap. The application was performed with the athletes in the supine semi-recumbent position.
  Interventions: Device: Cold Compression
- 10 Degree Cold Compression Group: Cold compression application was performed using Game Ready for 15 minutes. The target temperature was manually set to 10°C and the pressure to high compression (75 mm Hg). Pneumatic intermittent compression in a standard ∼3 min cycle was applied to both lower legs using a thigh wrap. The application was performed with the athletes in the supine semi-recumbent position.
  Interventions: Device: Cold Compression
- Passive Rest Control Group: The athletes rested passively in the supine semi-recumbent position for 15 minutes after the training.

INTERVENTIONS:
Device: Cold Compression — Cold compression was applied to the athletes with the Game Ready (Game Ready; Global, UK) device. The Game Ready (GR) device applies cooling to the tissue by continuous circulation of ice water with intermittent pneumatic compression. The GR consists of a sleeve that surrounds the affected tissue, a tank containing the ice water and a hose connecting the two. There are chambers inside the sleeve and the air pumped through these chambers and the broken ice pieces and water surround the tissue. The pressure settings are no compression (0 mmHg), low compression (5 to 15 mmHg), medium compression (5 to 50 mmHg) and high compression (5 to 75 mmHg). The ice water passes through the sleeve in 3-minute inflation and deflation cycles. The temperature of the water inside the device can be adjusted by adding ice and water. The temperature to be applied to the tissue is set with the screen on the device.
  Groups: 1 Degree Cold Compression Group; 10 Degree Cold Compression Group

SUMMARY:
Our study examining the effects of post-training cold compression on muscle oxygen saturation (MOS9), fatigue and jumping performance in professional male volleyball players.

DETAILED DESCRIPTION:
Volleyball is an intermittent sport consisting of short and high-intensity phases where players jump and change direction suddenly. Intense muscle use during training, intense match schedules, short preparation phases and double trainings applied during the day can cause athletes to lose performance and increase injury rates. The performance of the athlete during the season depends on the amount and distribution of the training load and the appropriate recovery intervention applied during the season. Therefore, appropriate recovery interventions for athletes, shortening the recovery period and increasing its quality are very important. Recovery is a process in which the athlete's fatigue after intense training or matches is eliminated, lactic acid in the muscle and blood is removed, energy stores are restored to their previous level and myoglobin oxygenation is provided. One of the parameters used to examine the effects of muscle damage after exercise and to follow recovery is oxygen saturation. It is known that oxygen saturation in the muscle decreases during exercise and increases in the following recovery process. Different interventions are recommended to optimize the recovery of athletes during the season. Cold applications are the most frequently preferred method due to their practicality and accessibility after training as a recovery intervention. Although it has been reported that cold applications have positive effects on fatigue and general perceptual well-being, their effects on acute performance parameters are controversial. In recent years, the use of cold compression applications in the recovery process after training has become widespread in clinics and sports clubs due to the fact that they allow two types of application and are portable and practical. Cold compression devices aim to reduce tissue temperature, reduce pain, control inflammation and accelerate venous return by applying cold and compression simultaneously. This is achieved by continuous circulation of ice water using intermittent pneumatic compression. There are many studies in the literature on the effects of cold applications on performance parameters (no effect or negative effect) and fatigue (reducing muscle pain and fatigue effects). However, the effect of cold compression on recovery at different temperatures has not been determined. Determining the degree of cold applied and the response received, as well as better identifying recovery interventions applied in professional sports environments and developing cold application protocols applied during the post-training recovery process, and investigating the effects of cold compression on fatigue, performance parameters and recovery parameters will contribute significantly to the literature. Therefore, the aim of our study is to examine the effects of different degrees of cold compression applied to professional male volleyball players compared to passive rest on muscle oxygen saturation, fatigue level and performance.

ELIGIBILITY:
Inclusion Criteria:

* Professional male volleyball player
* Performing 100-120 jumps in training (The number of jumps of the athletes in training was determined by Vert Classic (Model #JEM, Mayfonk Athletic, Fort Lauderdale, FL, USA).
* Body Mass Index (BMI) below 30 kg/m2
* Voluntary participation in the study

Exclusion Criteria:

* Smoking
* The presence of any neurological, rheumatologic or systemic disease
* Any injury or trauma to the quadriceps muscle and lower extremity in the last six months
* The athlete has exercised after training

Ages: 18 Years to 37 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men's
Study Population: Professional Men's Volleyball Players
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Muscle Oxygen Saturation Measurement | Muscle oxygen saturation measurements were taken before and immediately after training. Subsequently, the measurement was repeated after 15 minutes of passive rest or cold compression and 24 hours later at follow-up.
  Muscle oxygen saturation measurements of the athletes were performed with the MOXY device (Fortiori Design LLC., Minnesota, USA). The MOXY device sends 4 separate near infrared lights and works with a system that goes 12.5-25 mm deep into the skin and gives a numerical average of the amount of light reflected between the sensors. The infrared device, called near infrared spectroscopy (NIRS), measures total hemoglobin, oxygen saturation in capillaries and myoglobin saturation in the muscle. The electrodes are self-adhesive. The device has been shown to be a valid and reliable method for measuring muscle oxygenation (r=0.842-0.993, ICC: r=0.773-0.992). In the athletes in our study, superficial electrodes were placed midline on the quadriceps femoris muscle on the dominant side. Before placement, the electrode sites were shaved and cleaned with alcohol. All measurements were made at the same point and taken in the long sitting position.

SECONDARY OUTCOMES:
Fatigue Measurement | Fatigue measurements of the athletes were taken before and immediately after training. Subsequently, the measurement was repeated after 15 minutes of intervention and at follow-up after 24 hours.
  The degree of fatigue perceived by the athletes after training was recorded with the Modified Borg Scale (BORG CR-10 Scale). The scale developed by Borg consists of definitions that come to certain numbers. The scale was introduced to the athletes verbally. Fatigue was graded between 0 and 10 (0: None, 10: Maximum). The Modified Borg Scale has been shown to be a valid and reliable method for the assessment of fatigue.
Performance Measurement | The jump heights of the athletes were automatically recorded with the Vert Coach in the training just before the application and in the second training 24 hours later and were included in the evaluation form.
  Jump performance was evaluated with the Vert Coach (Mayfonk Athletic, Florida, USA). The device allows all athletes to measure and record jump height and number of jumps simultaneously during training or a match. It is frequently preferred due to its low cost and the fact that it does not require any extra measurement or effort for the performance evaluation of the athlete. The device measures 6×3×0.5 and has a motion-sensitive sensor on it. The sensor connected to the device is attached to the athlete's waist with an elastic belt. The sensor calculates the vertical displacement of each jump. The data is then transferred to a phone or tablet via bluetooth. The device has been shown to be a valid and reliable method of assessing vertical jump performance in volleyball players (r=0.75-0.97, ICC=0.97).

CONTACTS AND LOCATIONS:
Overall Officials: seval tamer, asist. prof, Principal Investigator — worker
Locations (1):
- Kutahya Health and Science University, Kütahya, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhambhani YN. Muscle oxygenation trends during dynamic exercise measured by near infrared spectroscopy. Can J Appl Physiol. 2004 Aug;29(4):504-23. doi: 10.1139/h04-033. PMID 15328597
- [Background] Alexander J, Jeffery J, Rhodes D. Recovery profiles of eccentric hamstring strength in response to cooling and compression. J Bodyw Mov Ther. 2021 Jul;27:9-15. doi: 10.1016/j.jbmt.2021.03.010. Epub 2021 Mar 28. PMID 34391318
- [Background] Chow GCC, Yam TTT, Chung JWY, Fong SSM. Effects of postexercise ice-water and room-temperature water immersion on the sensory organization of balance control and lower limb proprioception in amateur rugby players: A randomized controlled trial. Medicine (Baltimore). 2017 Feb;96(7):e6146. doi: 10.1097/MD.0000000000006146. PMID 28207546